CLINICAL TRIAL: NCT05361616
Title: Impact of Photobiomodulation on Pain During Orthodontic Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PBM Healing International Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00112179
Record Dates: First submitted 2021-07-13; First posted 2022-05-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Malocclusion; Orthodontic Treatment
Keywords: photobiomodulation; clear aligners; orthodontic pain
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PBM Ortho Active device (Active Comparator): PBM Ortho Active group will be given an active device.
  Interventions: Device: PBM Ortho
- PBM Ortho Sham (Sham Comparator): PBM Ortho Sham device group will be given a non-active device that will not emits light.
  Interventions: Device: PBM Ortho

INTERVENTIONS:
Device: PBM Ortho — The device will be used by the patients at home for one 8 minutes per day (4 minutes each upper and lower) for 7 days.

SUMMARY:
The objective of this study is to determine to effect of PBM Ortho, a photobiomodulation device, in adult patients undergoing clear aligners orthodontic treatment. We hypothesize that PBM Ortho will reduced the orthodontic associated pain in the clear aligner patients. This effect will be evaluated by recording the pain on visual analog scale given to the patients before the placement of clear aligners and collecting saliva.

DETAILED DESCRIPTION:
Pain associated with orthodontic treatment is one of the main causes of treatment discontinuation and patient non-cooperation. Several treatment modalities have been studied to alleviate orthodontic pain which includes pharmacological, mechanical, and behavioral approach. One potential treatment is the application of photobiomodulation (PBM) therapy which is a form of light therapy. The objective of this study is to determine to effect of PBM therapy in adult patients undergoing clear aligners orthodontic treatment. This effect will be evaluated by recording the pain on visual analog scale given to the patients before the placement of clear aligners and collecting saliva. The patients will be provided with active PBM Ortho device and sham PBM device (placebo, which will look similar to the active device) to use them at home for one 8 minutes application for 7 days (4 minutes per arch, upper or lower). The pain scale sheets will also be given to the patients to fill them every day for 7 days. The inflammatory protein associated with pain present in the saliva will be collected on Day 1 (24 hours after clear aligner treatment start), Day 4 (fourth day of treatment), and Day 7 (after 1 week from the treatment start). On the last visit, the device and pain scale sheets will be collected from the patients. If successful, this device therapy will reduce the orthodontic associated pain and improve patients' compliance and cooperation.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy male and female patients (age 20 to 65), i.e., do not suffer from systemic illness nor require medication during the saliva collection period.
* Permanent dentition, with Little's Irregularity Index (LII) of 2 mm or greater for the upper and lower arch.
* Orthodontic treatment using clear aligners via non-extraction therapy.
* Patient is available for follow-up visits.
* Patient is able and willing to comply with the requirements of this trial protocol.
* Non-smoker with no use of chewing tobacco.
* Good oral hygiene.
* Caries free.
* No sign of periodontal disease.

Exclusion Criteria:

* Systemic diseases
* Medication use for the past 6 months; specially use of anti-inflammatory (e.g., NSAIDs), antiviral, antibiotics.
* Smoking.
* Active dental caries.
* Any periodontal problem including bleeding, tooth mobility, bone loss, attachment loss, deep pockets.
* Sleep apnea and other airway pathologies.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-04-17 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Visual analog scale | Day 0: prior to seating first clear aligner tray
  Study endpoint for effectiveness in decreasing the pain perception during orthodontic tooth movement. Pain intensity will be scored between 0 (no pain) and 10 (worst imaginable pain) on the numeric scale. Pain intensity does not have a unit to describe. The pain intensity will be recorded in both groups at Day 0 (after the placement of the first composite attachments on the teeth but before the seating of the first clear aligner), and then every day for 7 consecutive days.
Visual analog scale | Day 1
  Study endpoint for effectiveness in decreasing the pain perception during orthodontic tooth movement. Pain intensity will be scored between 0 (no pain) and 10 (worst imaginable pain) on the numeric scale. Pain intensity does not have a unit to describe. The pain intensity will be recorded in both groups at Day 0 (after the placement of the first composite attachments on the teeth but before the seating of the first clear aligner), and then every day for 7 consecutive days.
Visual analog scale | Day 2
  Study endpoint for effectiveness in decreasing the pain perception during orthodontic tooth movement. Pain intensity will be scored between 0 (no pain) and 10 (worst imaginable pain) on the numeric scale. Pain intensity does not have a unit to describe. The pain intensity will be recorded in both groups at Day 0 (after the placement of the first composite attachments on the teeth but before the seating of the first clear aligner), and then every day for 7 consecutive days.
Visual analog scale | Day 3
  Study endpoint for effectiveness in decreasing the pain perception during orthodontic tooth movement. Pain intensity will be scored between 0 (no pain) and 10 (worst imaginable pain) on the numeric scale. Pain intensity does not have a unit to describe. The pain intensity will be recorded in both groups at Day 0 (after the placement of the first composite attachments on the teeth but before the seating of the first clear aligner), and then every day for 7 consecutive days.
Visual analog scale | Day 4
  Study endpoint for effectiveness in decreasing the pain perception during orthodontic tooth movement. Pain intensity will be scored between 0 (no pain) and 10 (worst imaginable pain) on the numeric scale. Pain intensity does not have a unit to describe. The pain intensity will be recorded in both groups at Day 0 (after the placement of the first composite attachments on the teeth but before the seating of the first clear aligner), and then every day for 7 consecutive days.
Visual analog scale | Day 5
  Study endpoint for effectiveness in decreasing the pain perception during orthodontic tooth movement. Pain intensity will be scored between 0 (no pain) and 10 (worst imaginable pain) on the numeric scale. Pain intensity does not have a unit to describe. The pain intensity will be recorded in both groups at Day 0 (after the placement of the first composite attachments on the teeth but before the seating of the first clear aligner), and then every day for 7 consecutive days.
Visual analog scale | Day 6
  Study endpoint for effectiveness in decreasing the pain perception during orthodontic tooth movement. Pain intensity will be scored between 0 (no pain) and 10 (worst imaginable pain) on the numeric scale. Pain intensity does not have a unit to describe. The pain intensity will be recorded in both groups at Day 0 (after the placement of the first composite attachments on the teeth but before the seating of the first clear aligner), and then every day for 7 consecutive days.
Visual analog scale | Day 7
  Study endpoint for effectiveness in decreasing the pain perception during orthodontic tooth movement. Pain intensity will be scored between 0 (no pain) and 10 (worst imaginable pain) on the numeric scale. Pain intensity does not have a unit to describe. The pain intensity will be recorded in both groups at Day 0 (after the placement of the first composite attachments on the teeth but before the seating of the first clear aligner), and then every day for 7 consecutive days.

SECONDARY OUTCOMES:
Saliva analysis | The saliva will be collected on Day 0
  2 ml of saliva samples will be obtained from all the patients enrolled in the study at Day 0, Day 1, Day 4 and Day 7 time points in 15-ml Falcon tubes. The samples will be immediately frozen and stored at -80°C refrigerator until assayed.
  Multiplex immunoassay will be used to analyze target proteins: cortisol, testosterone, alpha amylase, interleukin 1β (IL-1β), prostaglandin E2 (PGE2), receptor activator of nuclear factor kappa-B ligand (RANKL), nerve growth factor (NGF), brain derived neurotrophic factor (BDNF), substance P (SP), macrophage inflammatory protein-4 (MIP-4), matrix metalloproteinase-8 (MMP-8). ELISA kits for each target protein will be utilized to quantify the protein in the saliva and the unit will be according to the protocol provided in the kit.
Saliva analysis | The saliva will be collected on Day 1
  2 ml of saliva samples will be obtained from all the patients enrolled in the study at Day 0, Day 1, Day 4 and Day 7 time points in 15-ml Falcon tubes. The samples will be immediately frozen and stored at -80°C refrigerator until assayed.
  Multiplex immunoassay will be used to analyze target proteins: cortisol, testosterone, alpha amylase, interleukin 1β (IL-1β), prostaglandin E2 (PGE2), receptor activator of nuclear factor kappa-B ligand (RANKL), nerve growth factor (NGF), brain derived neurotrophic factor (BDNF), substance P (SP), macrophage inflammatory protein-4 (MIP-4), matrix metalloproteinase-8 (MMP-8). ELISA kits for each target protein will be utilized to quantify the protein in the saliva and the unit will be according to the protocol provided in the kit.
Saliva analysis | The saliva will be collected on Day 4
  2 ml of saliva samples will be obtained from all the patients enrolled in the study at Day 0, Day 1, Day 4 and Day 7 time points in 15-ml Falcon tubes. The samples will be immediately frozen and stored at -80°C refrigerator until assayed.
  Multiplex immunoassay will be used to analyze target proteins: cortisol, testosterone, alpha amylase, interleukin 1β (IL-1β), prostaglandin E2 (PGE2), receptor activator of nuclear factor kappa-B ligand (RANKL), nerve growth factor (NGF), brain derived neurotrophic factor (BDNF), substance P (SP), macrophage inflammatory protein-4 (MIP-4), matrix metalloproteinase-8 (MMP-8). ELISA kits for each target protein will be utilized to quantify the protein in the saliva and the unit will be according to the protocol provided in the kit.
Saliva analysis | The saliva will be collected on Day 7
  2 ml of saliva samples will be obtained from all the patients enrolled in the study at Day 0, Day 1, Day 4 and Day 7 time points in 15-ml Falcon tubes. The samples will be immediately frozen and stored at -80°C refrigerator until assayed.
  Multiplex immunoassay will be used to analyze target proteins: cortisol, testosterone, alpha amylase, interleukin 1β (IL-1β), prostaglandin E2 (PGE2), receptor activator of nuclear factor kappa-B ligand (RANKL), nerve growth factor (NGF), brain derived neurotrophic factor (BDNF), substance P (SP), macrophage inflammatory protein-4 (MIP-4), matrix metalloproteinase-8 (MMP-8). ELISA kits for each target protein will be utilized to quantify the protein in the saliva and the unit will be according to the protocol provided in the kit.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Sphinx Orthodontic, Edmonton, Alberta
  - Orthodontic Graduate Clinic, Kaye Clinic, University of Alberta, Edmonton, Alberta

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] White DW, Julien KC, Jacob H, Campbell PM, Buschang PH. Discomfort associated with Invisalign and traditional brackets: A randomized, prospective trial. Angle Orthod. 2017 Nov;87(6):801-808. doi: 10.2319/091416-687.1. Epub 2017 Jul 28. PMID 28753032
- [Background] Wiedel AP, Bondemark L. A randomized controlled trial of self-perceived pain, discomfort, and impairment of jaw function in children undergoing orthodontic treatment with fixed or removable appliances. Angle Orthod. 2016 Mar;86(2):324-30. doi: 10.2319/040215-219.1. Epub 2015 Jul 17. PMID 26185899
- [Background] Johal A, Fleming PS, Al Jawad FA. A prospective longitudinal controlled assessment of pain experience and oral health-related quality of life in adolescents undergoing fixed appliance treatment. Orthod Craniofac Res. 2014 Aug;17(3):178-86. doi: 10.1111/ocr.12044. Epub 2014 Apr 7. PMID 24703180
- [Background] Polat O, Karaman AI. Pain control during fixed orthodontic appliance therapy. Angle Orthod. 2005 Mar;75(2):214-9. doi: 10.1043/0003-3219(2005)0752.0.CO;2. PMID 15825785
- [Background] Long H, Wang Y, Jian F, Liao LN, Yang X, Lai WL. Current advances in orthodontic pain. Int J Oral Sci. 2016 Jun 30;8(2):67-75. doi: 10.1038/ijos.2016.24. PMID 27341389
- [Background] Panda S, Verma V, Sachan A, Singh K. Perception of pain due to various orthodontic procedures. Quintessence Int. 2015 Jul-Aug;46(7):603-9. doi: 10.3290/j.qi.a33933. PMID 25918756
- [Background] Baldini A, Nota A, Santariello C, Assi V, Ballanti F, Cozza P. Influence of activation protocol on perceived pain during rapid maxillary expansion. Angle Orthod. 2015 Nov;85(6):1015-20. doi: 10.2319/112114-833.1. Epub 2015 Mar 10. PMID 25757063
- [Background] Mangnall LA, Dietrich T, Scholey JM. A randomized controlled trial to assess the pain associated with the debond of orthodontic fixed appliances. J Orthod. 2013 Sep;40(3):188-96. doi: 10.1179/1465313313Y.0000000045. PMID 24009318
- [Background] Dray A. Inflammatory mediators of pain. Br J Anaesth. 1995 Aug;75(2):125-31. doi: 10.1093/bja/75.2.125. PMID 7577246
- [Background] Ren Y, Vissink A. Cytokines in crevicular fluid and orthodontic tooth movement. Eur J Oral Sci. 2008 Apr;116(2):89-97. doi: 10.1111/j.1600-0722.2007.00511.x. PMID 18353001
- [Background] Zeng M, Kou X, Yang R, Liu D, Wang X, Song Y, Zhang J, Yan Y, Liu F, He D, Gan Y, Zhou Y. Orthodontic Force Induces Systemic Inflammatory Monocyte Responses. J Dent Res. 2015 Sep;94(9):1295-302. doi: 10.1177/0022034515592868. Epub 2015 Jun 30. PMID 26130260
- [Background] Scott DA, Krauss J. Neutrophils in periodontal inflammation. Front Oral Biol. 2012;15:56-83. doi: 10.1159/000329672. Epub 2011 Nov 11. PMID 22142957
- [Background] Yan Y, Liu F, Kou X, Liu D, Yang R, Wang X, Song Y, He D, Gan Y, Zhou Y. T Cells Are Required for Orthodontic Tooth Movement. J Dent Res. 2015 Oct;94(10):1463-70. doi: 10.1177/0022034515595003. Epub 2015 Jul 17. PMID 26187644
- [Background] Topolski F, Moro A, Correr GM, Schimim SC. Optimal management of orthodontic pain. J Pain Res. 2018 Mar 16;11:589-598. doi: 10.2147/JPR.S127945. eCollection 2018. PMID 29588616
- [Background] Monk AB, Harrison JE, Worthington HV, Teague A. Pharmacological interventions for pain relief during orthodontic treatment. Cochrane Database Syst Rev. 2017 Nov 28;11(11):CD003976. doi: 10.1002/14651858.CD003976.pub2. PMID 29182798
- [Background] Ngan P, Kess B, Wilson S. Perception of discomfort by patients undergoing orthodontic treatment. Am J Orthod Dentofacial Orthop. 1989 Jul;96(1):47-53. doi: 10.1016/0889-5406(89)90228-x. PMID 2750720
- [Background] Fleming PS, Strydom H, Katsaros C, MacDonald L, Curatolo M, Fudalej P, Pandis N. Non-pharmacological interventions for alleviating pain during orthodontic treatment. Cochrane Database Syst Rev. 2016 Dec 23;12(12):CD010263. doi: 10.1002/14651858.CD010263.pub2. PMID 28009052
- [Background] Wu S, Chen Y, Zhang J, Chen W, Shao S, Shen H, Zhu L, Ye P, Svensson P, Wang K. Effect of low-level laser therapy on tooth-related pain and somatosensory function evoked by orthodontic treatment. Int J Oral Sci. 2018 Jul 2;10(3):22. doi: 10.1038/s41368-018-0023-0. PMID 29967411
- [Background] Al-Okla N, Bader D, Al-Mulla A, Ferguson D, Shaughnessy T. Effect of photobiomodulation on pain perception among orthodontic patients: a randomized clinical trial. J Clin Orthod. 2020 Feb;54(2):96-103. No abstract available. PMID 32554911
- [Background] Farias RD, Closs LQ, Miguens SA Jr. Evaluation of the use of low-level laser therapy in pain control in orthodontic patients: A randomized split-mouth clinical trial. Angle Orthod. 2016 Mar;86(2):193-8. doi: 10.2319/122214-933.1. Epub 2015 Jul 1. PMID 26132512
- [Background] Sfondrini MF, Vitale M, Pinheiro ALB, Gandini P, Sorrentino L, Iarussi UM, Scribante A. Photobiomodulation and Pain Reduction in Patients Requiring Orthodontic Band Application: Randomized Clinical Trial. Biomed Res Int. 2020 May 25;2020:7460938. doi: 10.1155/2020/7460938. eCollection 2020. PMID 32596367